CLINICAL TRIAL: NCT07385976
Title: The Role of Blood Perfusion in Cervical Cancer, Cervical Intraepithelial Neoplasm and Ovarian Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, MD, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 114237-F
Record Dates: First submitted 2026-01-13; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasm; Ovarian Cancer
Keywords: 3D power Doppler sonography; cervical vascularization and blood flow
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Ovarian Neoplasms | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- cervical cancer: cervical cancer patients
  Interventions: Diagnostic Test: Doppler ultrasound
- cervical intraepithelial neoplasm: cervical intraepithelial neoplasm patients
  Interventions: Diagnostic Test: Doppler ultrasound
- control: Gynecological patients without cervical disease
  Interventions: Diagnostic Test: Doppler ultrasound
- ovarian cancer: ovarian cancer patients
  Interventions: Diagnostic Test: Doppler ultrasound

INTERVENTIONS:
Diagnostic Test: Doppler ultrasound — 3D doppler ultrasound to measure VI, FI, VFI.

SUMMARY:
This study will elucidate the role of 3D transvaginal ultrasound in assessing (1) cervical vascularity and blood flow in patients with cervical cancer and cervical intraepithelial neoplasm, and (2) tumor vascularity and blood flow in patients with ovarian cancer.

DETAILED DESCRIPTION:
Patients and methods:

Women with cervical cancer, cervical intraepithelial neoplasm, ovarian cancer, or the control will be invited to particilate in this study.Then, 3D power Doppler Ultrasound will be performed to capture (1) the cervical volume, vascularity and blood perfusion, and (2) ovarian tumor vascularity and blood perfusion. The sonographic data will be correlated to clinical and pathological data.

ELIGIBILITY:
Inclusion Criteria:

* Regarding the topic "Hemoperfusion characteristics of cervical cancer and precancerous lesions, and the correlation between hemoperfusion and prognosis":

  1. Adult women who have had a normal cervical smear within the past three years and have no other gynecological cancers (control group).
  2. Adult women with cervical cancer or precancerous lesions.
* Regarding the topic "Correlation between hemoperfusion and prognosis of ovarian cancer":

  1. Adult women suspected of having ovarian cancer, fallopian tube cancer, or peritoneal cancer before surgery.

Exclusion Criteria:

* Regarding the topic "Hemoperfusion characteristics of cervical cancer and precancerous lesions of the cervix, and the correlation between hemoperfusion and prognosis":

  1. Patients who cannot cooperate with vaginal 3D ultrasound scans.
* Regarding the topic "Correlation between hemoperfusion and prognosis of ovarian cancer":

  1. Patients who cannot cooperate with vaginal or abdominal 3D ultrasound scans.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Women with cervical cancer, cervical intraepithelial neoplasm, ovarian cancer, and the disease-free control
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Vascularization-flow index | 3 years
  1. Compare the vascularization-flow index values between cervical cancer, cervical intraepithelial neoplasia and the control group.
  2. To assess whether vascularization-flow index is a predictor of progression-free survival in women with ovarian cancer

SECONDARY OUTCOMES:
Vascularization index | 3 years
  1. Compare the vascularization index values between cervical cancer, cervical intraepithelial neoplasia and the control group. 2. To assess whether vascularization index is a predictor of progression-free survival in women with ovarian cancer
Flow index | 3 years
  1. Compare the flow index values between cervical cancer, cervical intraepithelial neoplasia and the control group. 2. To assess whether flow index is a predictor of progression-free survival in women with ovarian cancer

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital,, New Taipei City, Banqiao
  - Far Eastern Memorial Hospital, New Taipei City

IPD SHARING:
Plan to Share IPD: No